CLINICAL TRIAL: NCT03599128
Title: Effect of Phenolic Acids on the Human Vasculature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 1717NRC
Record Dates: First submitted 2018-03-01; First posted 2018-07-26 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — phenolic acid; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 43.3 mg hydrolyzed green coffee extract (Experimental): hydrolyzed green coffee extract as interventions
  Interventions: Other: 43.3 mg hydrolyzed green coffee extract
- 86.6 mg hydrolyzed green coffee extract (Experimental): hydrolyzed green coffee extract as interventions
  Interventions: Other: 86.6 mg hydrolyzed green coffee extract
- 173 mg hydrolyzed green coffee extract (Experimental): hydrolyzed green coffee extract as interventions
  Interventions: Other: 173 mg hydrolyzed green coffee extract

INTERVENTIONS:
Other: 43.3 mg hydrolyzed green coffee extract — Reconstituted in water and given to subjects
  Other Names: Phenolic acid
  Arms: 43.3 mg hydrolyzed green coffee extract
Other: 86.6 mg hydrolyzed green coffee extract — Reconstituted in water and given to subjects
  Other Names: Phenolic acid
  Arms: 86.6 mg hydrolyzed green coffee extract
Other: 173 mg hydrolyzed green coffee extract — Reconstituted in water and given to subjects
  Other Names: Phenolic acid
  Arms: 173 mg hydrolyzed green coffee extract
Other: Placebo — Reconstituted in water and given to subjects
  Other Names: maltodextrin
  Arms: Placebo

SUMMARY:
This study evaluates effects of different doses of phenolic acids on healthy volunteers.

DETAILED DESCRIPTION:
It has been suggested that consumption of food rich in phenolic acids can help to improve vascular health, measured by flow mediated dilation (FMD).

ELIGIBILITY:
Inclusion Criteria:

* Male or postmenopausal female healthy volunteers aged 45-65 years old
* Willing and able to sign written informed consent prior to trial entry
* Healthy as determined by the medical history and physical examination

Exclusion Criteria:

* Premenopausal women
* Current smokers
* Abnormal blood pressure as defined as follow: systolic <90 or >140 mmHg and diastolic <60 or >90 mmHg
* Regular consumption of cholesterol-lowering medication
* Regular consumption of antihypertensive medication
* Regular consumption of any vasoactive medication that cannot be discontinued for at least 4 half-lives before the FMD assessment
* Any food allergies
* Any intakes of multivitamin-tablets and other supplemental compounds 10 days before the study start and throughout the study
* Inability to refrain from coffee/tea and alcohol consumption for 12 h prior to study visits
* Acute or chronic major psychiatric illness or other major illness that in the opinion of the investigator would make the subjects' participation in the study unsafe or prevent them from fully complying with the study procedures
* Body mass index (BMI) outside 18-32 kg/m2 range

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Efficacy by oral administration of phenolic acid in improving endothelial function | 6 hours
  Average change from baseline in %FMD at any time point post treatment. Responses will be calculated as the percentage change in brachial artery diameter from baseline.

SECONDARY OUTCOMES:
AUC(Area Under Curve) of the concentration/time curve | 6 hours
  link between endothelial function improvement in healthy subjects and plasma concentration of phenolic acids
Tmax | 6 hours
  link between endothelial function improvement in healthy subjects and plasma concentration of phenolic acids
Elimination half-life | 6 hours
  link between endothelial function improvement in healthy subjects and plasma concentration of phenolic acids

OTHER OUTCOMES:
Blood concentrations in plasma. | 6 hours
  Blood concentrations in plasma.
To investigate safety of investigational products: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year.
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Tan, Study Chair — Société des Produits Nestlé (SPN)
Locations (1):
- University of Western Australia, Crawley, Perth, Australia

IPD SHARING:
Plan to Share IPD: Undecided